CLINICAL TRIAL: NCT01082939
Title: A Phase II Study of Cyclophosphamide, Fludarabine, Alemtuzumab, and Rituximab (CFAR) in Previously Treated Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Cyclophosphamide, Fludarabine, Alemtuzumab, and Rituximab (CFAR) for Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM02-593
Record Dates: First submitted 2010-03-05; First posted 2010-03-09 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; Refractory CLL; CFAR; Alemtuzumab; Campath-1H; Campath; Cyclophosphamide; Cytoxan; Neosar; Fludarabine; Fludara; Fludarabine Phosphate; Rituximab; Rituxan; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CFAR (Experimental): CFAR: Cyclophosphamide 250 mg/m^2/day intravenous (IV) Days 3-5, Fludarabine 25 mg/m^2/day IV Days 3-5, Alemtuzumab 30 mg IV Days 1, 3 and 5 over 2-4 hours, repeated every four weeks for a total of 6 planned cycles, and Rituximab Cycle 1 (Week 1): 375 mg/m^2/day IV Day 2 over 4- 6 hours, Cycle 2 - 6 (Week 1): 500 mg/m^2/day IV Day 2 over 4- 6 hours.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Alemtuzumab; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2/day IV on Days 3-5; repeated every four weeks for a total of 6 planned cycles.
  Other Names: Fludara; Fludarabine Phosphate
Drug: Cyclophosphamide — 250 mg/m^2/day IV on Days 3-5; repeated every four weeks for a total of 6 planned cycles.
  Other Names: Cytoxan; Neosar
Drug: Alemtuzumab — 30 mg IV on Days 1, 3 and 5 over 2-4 hours; repeated every four weeks for a total of 6 planned cycles.
  Other Names: Campath-1h; Campath
Drug: Rituximab — Cycle 1 (Week 1): 375 mg/m^2/day IV on Day 2 over 4- 6 hours
  Cycle 2 - 6 (Week 1): 500 mg/m^2/day IV on Day 2 over 4- 6 hours
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if the combination of fludarabine, cyclophosphamide, alemtuzumab, and rituximab is effective in treating chronic lymphocytic leukemia in patients who have already been treated with chemotherapy.

Primary Objectives:

Evaluate the therapeutic efficacy, including the complete remission (CR), nodular partial remission (NPR), and partial remission (PR) rates (overall response) of combined cyclophosphamide, fludarabine, alemtuzumab, and rituximab (CFAR) in previously treated patients with Chronic Lymphocytic Leukemia (CLL).

Second Objectives:

* Assess the toxicity profile of CFAR in previously treated patients with CLL.
* Monitor for infection and determine incidence and etiology of infection including cytomegalovirus in patients treated with CFAR.
* Evaluate molecular remission by polymerase chain reaction (PCR) for the clonal immunoglobulin heavy chain variable gene in responding patients treated with CFAR.
* Assess immune parameters, including pretreatment, during treatment, and post-treatment blood T-cell counts and subset distribution and serum immunoglobulin levels in patients treated with CFAR.

DETAILED DESCRIPTION:
Fludarabine is a chemotherapy drug that is approved for the treatment of CLL. Cyclophosphamide is also a chemotherapy drug that is commonly used in the treatment of CLL. Rituximab and alemtuzumab are special proteins that specifically target and attach to proteins on leukemia cells. These targeted proteins may also be present on normal blood cells. When these drugs bind to the proteins on leukemia cells, they may help to stop or slow the growth of the disease. The combination of fludarabine, cyclophosphamide and rituximab has been used in the treatment of CLL. The purpose of this study is to determine if there is added benefit with the addition of alemtuzumab to this combination.

Before treatment starts, you will have a complete physical exam, including blood tests (about 3 tablespoons). You may have either a chest x-ray or a computed tomography (CT) scan if your doctor feel this is necessary. If you have not had a bone marrow sample collected in the past 4 months, you will have a bone marrow sample collected at this time. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anaesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood pregnancy test.

During the study, you will have up to 6 "cycles" of treatment. A cycle is made up of treatment with the study drugs for 5 days in a row, then around 31/2 weeks (23 days) of no treatment with the study drugs. On Days 1, 3, and 5 of each cycle you will receive alemtuzumab through a needle in a vein. On Day 2 of each cycle you will receive rituximab through a needle in a vein. Cyclophosphamide and fludarabine will be given separately on Days 3, 4, and 5 of each cycle through a needle in a vein. In addition to the study drugs, you may also be given fluids by vein. The combination treatment will be repeated every 4 weeks (one cycle) for a total of up to 6 cycles. This treatment will be given on an outpatient basis. The injections for each daily treatment visit should take less than 6 hours.

You will receive acetaminophen (Tylenol) by mouth and diphenhydramine hydrochloride (Benadryl) by mouth or vein 30 - 60 minutes before each dose of rituximab and alemtuzumab. You will also receive hydrocortisone (a steroid) by vein before each dose of alemtuzumab. These drugs will be used to help decrease side effects. If side effects occur during a treatment, the doses of the drugs may be adjusted (up or down) until the symptoms are gone. Also, if you experience side effects during treatment, you must stay in the clinic for 2 hours after the drug is given to be observed.

If you begin to experience side effects due to treatment, the dose(s) of the drug(s) may be lowered or the treatment may be temporarily stopped until the symptoms are gone.

During the treatment and for two months after completion of treatment you will need to take prophylactic antibiotics to prevent you from developing infection. Trimethoprim/sulfamethoxazole (Bactrim DS) is a sulfa-drug and you will be given this to prevent a type of pneumonia called PCP pneumonia. If you are allergic to sulfa drugs, an equivalent antibiotic will be given. You will take Valtrex to prevent virus reactivation including herpes. If you are allergic to Valtrex, an equivalent antibiotic will be given. You may receive an additional antibiotic to suppress another virus, cytomegalovirus called Valcyte. You may also take allopurinol for the first week of the first course of treatment. This will help prevent kidney damage from rapid destruction of your leukemia cells.

During the first cycle of treatment, you will have blood drawn (about 2 tablespoons) for blood tests once a week. Then, these blood tests will be repeated before the start of each additional cycle (every 4 weeks).

After 3 cycles of treatment, you will have a physical exam and blood tests (about 2 tablespoons). You may also have either an x-ray or a CT scan. You will have another bone marrow sample collected. These tests will be used to see if the disease is responding to treatment. If it is found that the disease is not responding to treatment after the first 3 cycles of therapy, you will be taken off the study and your doctor will discuss other treatment options with you. If it is found that the disease is responding to treatment, another 3 cycles (12 weeks) of treatment will be given (6 cycles total). During these additional 3 cycles of therapy, you will have blood drawn (about 2 tablespoons) once a week for routine blood tests.

After 6 cycles of treatment, you will have a physical exam and have around 2 tablespoons of blood drawn for routine blood tests.

Around 3-6 months after you receive your last treatment cycle, you will have a physical exam and blood tests (about 2 tablespoons). After that, you will have a physical examination and blood tests (about 2 tablespoons) every 6 months for the next 2 years. If your disease returns or if you start on more treatment, you will not need to return for these visits. However, you should inform the study doctor/staff that you are receiving other treatment.

If at any time during the study the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

This is an investigational study. All of the drugs used in the study are FDA approved and commercially available. As many as 80 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have been diagnosed with CLL by immunophenotyping and flow cytometry analysis of blood or bone marrow demonstrating a monoclonal population of CD5 and CD19 positive cells.
2. All patient must have been previously treated with chemotherapy.
3. All patients with Rai stage III-IV are eligible for treatment with this protocol. - OR - All patients with Rai stage 0-II who meet one or more indication for treatment as defined by the NCI-sponsored Working Group are eligible for treatment with this protocol.
4. All patients must have a Zubrod performance status of 0-3.
5. All patients must have adequate renal and hepatic function (serum creatinine <2mg/dL; total bilirubin <2.5mg/dL). Patients with renal or liver dysfunction due to organ infiltration by lymphocytes may be eligible after discussion with the Principle Investigator and appropriate dose adjustment considered.
6. Patients may not receive concurrent chemotherapy, radiotherapy, or immunotherapy. Localized radiotherapy to an area not compromising bone marrow function does not apply, nor do hematopoietic growth factors such as erythropoietin, Granulocyte colony-stimulating factor (G-CSF or GCSF, GM-CSF etc).
7. Patients must not have untreated or uncontrolled life-threatening infection.
8. Patients must sign informed consent.

Exclusion Criteria:

1. None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PhD, BS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 12/6/02- 9/22/06; all participants were registered at The University of Texas M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | CFAR
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CFAR
Number analyzed (Participants) | 80
Age Continuous [Median (Full Range); unit: years] | 59.5 [39 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 66
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Overall Response
Description: Overall (OR) is the total number of participants with any response: Complete remission (CR), is defined as > 30% lymphocytes in the bone marrow, recovery of blood counts and no clinical symptoms; Nodular partial remission (NPR), is the same as CR but with nodules; Partial remission (PR) is > 50% decrease of clinical symptoms from baseline and recovery from blood counts.
Time Frame: 6 cycles of treatment (28 days per cycle)
Measure: Number; unit: Participants
Arm/Group | CFAR
Number analyzed (Participants) | 80
Participants
  Complete remission (CR) | 23
  Nodular partial remission (NPR) | 3
  Partial remission (PR) | 26

ADVERSE EVENTS:
Time Frame: 9 years
Arm/Group | CFAR
Serious Adverse Events (participants affected / at risk) | 35/80
Other Adverse Events (participants affected / at risk) | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CFAR (N=80)
Infection (Infections and infestations) | 22 (33)
Mucositis (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
fever (General disorders) | 10 (11)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Allergic Reaction (General disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Death (General disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CFAR (N=80)
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 4 (4)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Pure red cell aplasia (Blood and lymphatic system disorders) | 3 (3)
Cytomegalovirus Reactivation (Immune system disorders) | 9 (9)
drug reaction (General disorders) | 40 (40)
rash (Skin and subcutaneous tissue disorders) | 32 (32)
Nausea (Gastrointestinal disorders) | 33 (33)
Diarrhea (Gastrointestinal disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes